CLINICAL TRIAL: NCT02770781
Title: Feasibility Study of the Addition of a Personal Trainer to the Post-Treatment Regimen of Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Van Londen, Gijsberta, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-064
Record Dates: First submitted 2015-06-03; First posted 2016-05-12 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: survivors; physical fitness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Personal Trainer (Experimental): All subjects will meet a set amount of times with a personal trainer over the course of the study to participate in an exercise regimen.
  Interventions: Other: Exercise regimen

INTERVENTIONS:
Other: Exercise regimen — Subjects will receive a personal exercise regimen based on their health history and individual capability.

SUMMARY:
The purpose is to examine the feasibility and preliminary effectiveness of the role of a personal trainer for non-metastatic breast cancer survivors to improve physical activity and well-being (in terms of quality of life).

DETAILED DESCRIPTION:
After breast cancer treatment, many women are faced with effects of treatment such as changes in appearance, fatigue, and reduced quality of life as compared to the pre-disease state. An intervention to increase physical activity may be helpful to improve well-being and outcomes for women treated for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Post active breast cancer therapy (e.g. surgery and/or chemotherapy and/or radiation therapy), but may still be undergoing maintenance cancer therapy.
* Free of macro-metastatic disease
* Sedentary pre-cancer diagnosis: Those individuals not participating in a regular exercise program or not meeting the minimal physical activity recommendations from the General Surgeon which is accumulating 30 minutes or more of moderate physical activity on most days of the week
* Ability to provide informed consent
* Ability to provide a written physician's clearance
* Patients must be new to the Survivorship Clinic (within first 12 months).

Exclusion Criteria:

* Medical conditions that would preclude participation in a weight-training program.
* Those who plan on relocating outside the Greater Pittsburgh Area in the next 3 months of intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-10; Primary Completion 2018-04 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Study recruitment ability | Baseline through ~ 6 months of follow-up.
  Pilot study

SECONDARY OUTCOMES:
Physical fitness | Baseline through ~ 6 months of follow-up.
  Measured by pedometer.
Change in Paffenberger Exercise habits questionnaire | Baseline and ~ 6 months
  This questionnaire asks about exercise habits.
Change in physical activity self-efficacy questionnaire | Baseline and ~ 6 months
  This questionnaire will measure a person's perceived competence to engage in an activity
Functional Assessment of Cancer Therapy - Endocrine Symptoms | Baseline and ~ 6 months
  This is a quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: G van Londen, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Department of Medicine., Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qiao Y, van Londen GJ, Brufsky JW, Poppenberg JT, Cohen RW, Boudreau RM, Glynn NW. Perceived physical fatigability improves after an exercise intervention among breast cancer survivors: a randomized clinical trial. Breast Cancer. 2022 Jan;29(1):30-37. doi: 10.1007/s12282-021-01278-1. Epub 2021 Jul 30. PMID 34328623